CLINICAL TRIAL: NCT06379412
Title: A Cross-sectional Study on the Association of Peptidoglycan Fragments Derived From Gut Microbiota With Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhujianghmy
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Colorectal Cancer(CRC): People who are diagnosed with CRC by colonoscopy and pathological biopsy
  Interventions: Other: observational study, no intervention
- Colorectal adenoma(CRA): People who are diagnosed with CRA by colonoscopy and pathological biopsy
  Interventions: Other: observational study, no intervention
- Colorectal polyp(CRP): People who are diagnosed with CRP by colonoscopy and pathological biopsy
  Interventions: Other: observational study, no intervention
- Healthy: People who have no obvious abnormality in the whole colon
  Interventions: Other: observational study, no intervention

INTERVENTIONS:
Other: observational study, no intervention — observational study, no intervention

SUMMARY:
The goal of this observational study is to explore the association of peptidoglycan fragments derived from gut microbiota with colorectal cancer (CRC). The main question it aims to answer is: Are peptidoglycan fragments from the gut microbiota associated with the progression of colorectal cancer? Participants will provide biological specimens (blood, feces, colon tissue obtained during surgery)

DETAILED DESCRIPTION:
To explore whether peptidoglycan fragments can be used as screening or diagnostic indicators for colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* People who underwent total colonoscopy in gastroenteroscopy room.
* People who agree to participate in this study and are willing to sign informed consent.

Exclusion Criteria:

* Previous diagnosis of malignant tumors other than colorectal cancer.
* Received any of the following drug treatments within 1 month before sample collection: ① Drugs used for the treatment of colorectal diseases; ② Antibiotics; ③probiotics; ④ Laxatives.
* Patients with a family history of colorectal cancer.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Meet eligibility criteria
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
HPLC-MS/MS was used to detect peptidoglycan fragment content in biological specimens of 200 participants | baseline (before treatment)
  The content of peptidoglycan fragments was detected by HPLC-MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: He Xiaolong, Professor, Study Director — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China